CLINICAL TRIAL: NCT04672421
Title: A Comparative, Evaluator Blinded, Randomized, Multi-center Study to Evaluate the Efficacy and Safety of Medicurtain® in Patients With Total Laparoscopic Hysterectomy
Brief Title: The Efficacy and Safety of Medicurtain® in Patients With Total Laparoscopic Hysterectomy (Pivotal Study)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shin Poong Pharmaceutical Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: UMT2009-SP-ASMC-0301
Record Dates: First submitted 2020-11-29; First posted 2020-12-17 (Actual); Last update posted 2021-09-29 (Actual); Status verified 2021-09

CONDITIONS: Laparoscopy; Tissue Adhesion, Surgery-Induced; Leiomyoma of the Uterine Body
Keywords: Medicurtain®; Sodium hyaluronate; Hydroxyethylstarch; Anti-adhesion barrier
MeSH Terms: conditions — Tissue Adhesions; Myofibroma

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Evaluator-blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Medicurtain® (Experimental): Treat Medicurtain® 5ml prefilled syringe after laparoscopic surgery
  Interventions: Device: Medicurtain®
- Placebo (Sham Comparator): laparoscopic surgery
  Interventions: Device: Placebo

INTERVENTIONS:
Device: Medicurtain® — Anti-adhesion barrier (Medicurtain® 5ml prefilled syringe after laparoscopic surgery)
  Arms: Medicurtain®
Device: Placebo — No device after laparoscopic surgery
  Arms: Placebo

SUMMARY:
This study was designed to assess the safety and efficacy of MEDICURTAIN. Patients who underwent total laparoscopic hysterectomy were randomly assigned either into Medicurtain® treatment group or non-treatment control group. Adhesion formations at 8 weeks after the index surgery were compared between the two groups by using the well-defined grade scale and image recording.

DETAILED DESCRIPTION:
This study was designed as multi-center, randomized, evaluator-blinded, comparative study. Subjects were woman between 20~80 years of age reserved with total laparoscopic hysterectomy. Subject screening was conducted for the subject who signed an informed consent form. Subjects who met the inclusion criteria were randomly assigned into either treatment (Medicurtain®) or control group.

Each subject visit clinic for follow-up examination 1week (Visit 2) and 8 weeks (Visit 3) after the index surgery and before the visit subjects were received phone calls. Since the target population was the patient who scheduled elective total laparoscopic hysterectomy, subjects who met the inclusion/exclusion criteria after the examination for the surgery signed on the informed consent at Visit 1 (Baseline: 0 day) and randomly assigned either into the treatment and control group.

At visit 2 (1week±2days), 1week after the index surgery adverse events and general health were examined. At visit 3 (8week±5days), 8 weeks after the index surgery, the investigator inserted endoscope into abdominal cavity and took video clip and still images. If it was necessary, adhesion was removed surgically. An independent evaluator evaluated the records and graded the adhesion rate and its severity according to the grading system. If it was difficult to collect images with endoscope, the investigators recorded his observation for statistical analysis.

The investigator inserted endoscope into abdominal cavity and took video clip and still images at 8weeks after total laparoscopic hysterectomy to evaluate the adhesion formation and its grade. An independent evaluator evaluated the records and graded the adhesion rate and its severity according to the grading system. If it was difficult to collect images with endoscope, the investigators recorded his observation for statistical analysis. The adhesion grading system was proposed by American Fertility Society (AFS) in 1988, grades adhesion with Grade 0, Grade 1, Grade2 and Grade 3. Grade 0 means there is no adhesion formation, Grade 1~Grade 3 means there is adhesion formed, severity increases with the grade. Adhesion rate and grade were evaluated between the treatment and control groups suing Grade 0~3 scales.

General safety of the study device was evaluated based on the adverse event rate, laboratory tests, ECG test. The laboratory tests were conducted before and after the index surgery to evaluate whether the device cause toxicity such as hepatic and renal toxicity for safety evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Woman who is between 20~80 years of age.
* Woman who is reserved with total laparoscopic hysterectomy like:

  * Malignant neoplasm of cervix
  * Malignant neoplasm of uterine body
  * Unspecified malignant neoplasm of cervical region
  * Other and unspecified malignant neoplasm of the female reproductive system
  * Carcinoma in situ of the cervix
  * Other and unspecified carcinoma in situ of the reproductive system Leiomyoma of the uterus
  * Other benign neoplasms of uterus
  * Neoplasm of uncertain behavior of uterus
  * Endometriosis
  * Polyp of corpus uteri
  * Other noninflammatory disorders of uterus, except cervix
  * Cervical dysplasia
  * Congenital malformations of uterus and cervix
  * Injury of uterus
* Woman who signed and informed consent.

Exclusion Criteria:

* Presence of tumor or inflammatory disease in other organs after the laparoscopy or laparoscopic surgery
* Subjects with a history of open surgery or laparoscopic surgery
* Subject who is not eligible for anesthesia or re-operation due to other disease confirmed by investigator
* Subject who is not eligible for re-operation or laparoscopy after laparoscopic surgery
* Subjects using coagulant and subjects with lymphoid disease
* Diabetic subjects administrating oral or parenteral glucose-lowering drugs
* Patients with autoimmune diseases or immune disorders
* Liver disease or kidney disease, surgical subjects including open surgery of gastrointestinal or urinary system
* Subjects judged as inadequate by investigator

Ages: 20 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 107 (Actual)
Dates: Start 2011-04-18 (Actual); Primary Completion 2012-05-09 (Actual); Study Completion 2012-05-09 (Actual)

PRIMARY OUTCOMES:
Comparison of the adhesion rate between the groups | 8 weeks after surgery
  Adhesion rate = (number of subjects who developed adhesion in a group)/ (Total number of subjects for each group)

SECONDARY OUTCOMES:
Comparison of adhesion grade based on the severity between the groups | 8 weeks after surgery
  Adhesive grade evaluation standards are classified into Grade 0(None), Grade 1(Mild), Grade 2(Moderate), Grade 3(Severe).

OTHER OUTCOMES:
The incidence rate of adverse events | follow up to 8 weeks
  Safety and tolerability by collecting adverse events (AEs)
The incidence rate of adverse device event | follow up to 8 weeks
  Safety and tolerability by collecting adverse device event (ADEs)
The incidence rate of serious adverse events | follow up to 8 weeks
  Safety and tolerability by collecting serious adverse events (SAEs)
QT interval on a 12-lead electrocardiogram (ECG) tracing | follow up to 8 weeks
  Change From baseline in QT Interval

CONTACTS AND LOCATIONS:
Overall Officials: Young-Tak Kim, MD, PhD, Principal Investigator — Asan Medical Center, Seoul Asan Medical Center Gil, Songpa-gu, Seoul, Korea; Tae Jin Kim, MD, PhD, Principal Investigator — Cheil General Hospital & Women's Healthcare Center, 1-19 Mukjeong-dong, Jung-gu, Seoul, Korea; Yong-Il Kwon, MD, PhD, Principal Investigator — Kangdong Sacred Heart Hospital, (Gil 1dong445) 150, Seongnae-gil, Gwangsan-gu, Gwangju, Korea
Locations (1):
- Asan Medical Center, Seoul, Seoul Asan Medical Center Gil, Songpa-gu, South Korea

IPD SHARING:
Plan to Share IPD: No